CLINICAL TRIAL: NCT00491140
Title: Retrospective Study Assessing Molecular Features Predicting Response or Resistance to Cetuximab Therapy in Metastatic Colorectal Cancer Patients
Brief Title: Retrospective Study Assessing Molecular Features Predicting Response to Cetuximab
Status: Completed | Type: Observational
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Dr. Armando Santoro, Istituto Clinico Humanitas
Other Study IDs: ICH n. 380
Record Dates: First submitted 2007-06-22; First posted 2007-06-25 (Estimated); Last update posted 2008-10-01 (Estimated); Status verified 2008-09

CONDITIONS: Colorectal Neoplasms
Keywords: EGFR; KRAS; BRAF; MET; IGFR1
MeSH Terms: conditions — Colorectal Neoplasms | interventions — In Situ Hybridization, Fluorescence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Paraffine embedded tumor sections
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Observation: Colorectal cancer patients
  Interventions: Genetic: Gene mutations analysis and FISH

INTERVENTIONS:
Genetic: Gene mutations analysis and FISH — FISH and mutation analysis of multiple genes

SUMMARY:
The primary objective is to identify molecular features predicting response or resistance to cetuximab

DETAILED DESCRIPTION:
Secondary objective is to investigate association of genomic status of EGFR and HER-2 genes with clinical outcome, including objective response, time to progression and survival

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of colorectal cancer with available tumor tissue and clinical data; presence of at least one measurable lesion.

Exclusion Criteria:

* Less than 3 weeks after completion of previous radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Colorectal cancer patients treated with Cetuximab
Sampling Method: Non-Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2006-12; Primary Completion 2007-05 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Association of different biomarkers with Cetuximab sensitivity | Assessment every two months

SECONDARY OUTCOMES:
Association of different biomarkers with time to progression and survival | At the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Armando Santoro, MD, Study Director — Istituto Clinico Humanitas
Locations (1):
- Istituto Clinico Humanitas, Rozzano, Milan, Italy

REFERENCES:
- [Background] Chung KY, Shia J, Kemeny NE, Shah M, Schwartz GK, Tse A, Hamilton A, Pan D, Schrag D, Schwartz L, Klimstra DS, Fridman D, Kelsen DP, Saltz LB. Cetuximab shows activity in colorectal cancer patients with tumors that do not express the epidermal growth factor receptor by immunohistochemistry. J Clin Oncol. 2005 Mar 20;23(9):1803-10. doi: 10.1200/JCO.2005.08.037. Epub 2005 Jan 27. PMID 15677699